CLINICAL TRIAL: NCT00742963
Title: A Phase 1/2, Multicenter, Dose-Escalation Study to Determine the Safety, Efficacy and Pharmacokinetics of TH-302 in Combination With Doxorubicin in Patients With Advanced Soft Tissue Sarcoma
Brief Title: Dose-Escalation Study of TH-302 in Combination With Doxorubicin to Treat Patients With Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmunoGenesis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-403
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Soft Tissue Sarcoma
Keywords: TH-302; Advanced Soft Tissue Sarcoma; Doxorubicin; Phase 1/2
MeSH Terms: conditions — Sarcoma | interventions — TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 75 mg/m2 of Doxorubicin administered by bolus injection starting on Day 1 of a 21-day cycle.
  Interventions: Drug: TH-302

INTERVENTIONS:
Drug: TH-302 — TH-302 will be administered by IV infusion over 30-60 minutes on Days 1 and 8 of a 21-day cycle.
  Dose escalation dose levels:
  Dose level -1 (if needed): 180 mg/m2 Starting dose: 240 mg/m2

SUMMARY:
The purpose of this study is to determine whether TH-302 in combination with Doxorubicin is safe and effective in the treatment of Advanced Soft Tissue Sarcoma.

DETAILED DESCRIPTION:
A broad range of tumors have been shown to contain significant numbers of hypoxic cells and hypoxia has been shown to be associated with a poor prognosis and an increase in resistance to chemotherapy and radiotherapy (Brizel 1997, Vaupel 2007, Shannon 2003).

It is likely that an agent that could effectively target hypoxic regions in tumors would improve efficacy when combined with standard chemotherapy or radiotherapy. TH-302 is activated at lower oxygen concentrations than other bioreductive prodrugs (Duan 2008) and tirapazamine, a hypoxic cytotoxin that has been extensively studied in both preclinical and clinical studies. This should result in an improved therapeutic ratio (tumor vs normal tissue toxicity) as compared with other bioreductive agents. Because TH-302 is expected to be minimally toxic to aerobic cancer cells, optimal efficacy would be expected when TH-302 is combined with treatments that are most effective under aerobic conditions such as radiotherapy and cytotoxic chemotherapy. Preclinical data have shown at least additive efficacy when TH-302 is combined with chemotherapy. In order to minimize the risk of additive toxicity, TH-302 is not being evaluated in combination with alkylating agents. The study will enroll subjects with advanced soft tissue sarcoma. These tumors have evidence supporting the presence of hypoxia based on pO2 histography, F-MISO and gene expression profiling (Vaupel 2007, Francis 2007, Rajendran 2003).

ELIGIBILITY:
Inclusion Criteria

All Subjects:

* At least 18 years of age
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* Pathologically confirmed diagnosis of soft tissue sarcoma of the following subtypes:
* Synovial sarcoma
* High grade fibrosarcoma
* Unclassified, undifferentiated sarcoma
* Liposarcoma
* Leiomyosarcoma (excluding GIST)
* Angiosarcoma (excluding Kaposi's sarcoma)
* Pleomorphic sarcoma/malignant fibrous histiocytoma
* Locally advanced unresectable or metastatic disease with no standard curative therapy available and for whom treatment with single agent doxorubicin is considered appropriate; subjects in the dose escalation cohorts must have progressed since their most recent systemic therapy
* Recovered from reversible toxicities of prior therapy
* Evaluable disease by RECIST criteria (at least one target or non-target lesion for dose escalation cohorts; at least 1 target lesion for dose expansion cohort)
* ECOG performance status of 0 or 1
* Life expectancy of at least 3 months
* Acceptable liver function:
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN
* Acceptable renal function:
* Serum creatinine within normal limits
* Acceptable hematologic status (without hematologic support):
* ANC ≥ 1500 cells/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9.0 g/dL
* Acceptable cardiac function:
* Normal 12-lead ECG (clinically insignificant abnormalities permitted)
* LVEF normal by MUGA or echocardiogram
* Urinalysis: No clinically significant abnormalities
* All women of childbearing potential must have a negative serum pregnancy test and all subjects must agree to use effective means of contraception (surgical sterilization or the use or barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose

Exclusion Criteria

Prior therapy:

* Dose escalation cohort: Prior treatment with more than 2 myelosuppressive cytotoxic chemotherapy regimens
* Expanded cohort: Prior systemic therapy for advanced disease (neoadjuvant and adjuvant permitted)
* Low grade tumors according to standard grading systems (eg AJCC Grade 1 and 2)
* Prior therapy with ifosfamide or cyclophosphamide
* Prior therapy with an anthracycline or anthracenedione
* Prior mediastinal/cardiac radiotherapy
* Current use of drugs with known cardiotoxicity or known interactions with doxorubicin (see product label)
* Anticancer treatment with radiation therapy, chemotherapy, targeted therapies (erlotinib, lapatinib, etc.), immunotherapy, hormones or other antitumor therapies within 4 weeks prior to study entry (6 weeks for nitrosoureas or mitomycin C)
* Significant cardiac dysfunction:
* Any history of congestive heart failure
* Any history of transmural myocardial infarction
* Uncontrolled arrhythmias within the past 6 months
* Angina pectoris requiring antianginal medication within the past 6 months
* Clinically significant valvular heart disease
* Poorly controlled hypertension within the last 6 months
* Seizure disorders requiring anticonvulsant therapy
* Known brain metastases (unless previously treated and well controlled for a period of ≥ 3 months) Previously treated malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years
* Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation <90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause normal tissue hypoxia
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Prior therapy with an hypoxic cytotoxin
* Subjects who participated in an investigational drug or device study within 28 days prior to study entry
* Known infection with HIV, hepatitis B, or hepatitis C
* Subjects who have exhibited allergic reactions to a structural compound, biological agent, or formulation (containing solutol and/or propylene glycol) similar to TH-302
* Females who are pregnant or breast-feeding
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Unwillingness or inability to comply with the study protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-08; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Ganjoo, MD, Principal Investigator — Stanford University
Locations (9):
- United States (9):
  - Arizona Cancer Center, Tucson, Arizona
  - Sarcoma Oncology Center, Santa Monica, California
  - Stanford University, Stanford, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washingon University Siteman Cancer Center, St Louis, Missouri
  - Mary Crowley Cancer Research Centers, Dallas, Texas

REFERENCES:
- See also: Threshold Pharmaceuticals Company Website — http://www.thresholdpharm.com

RESULTS

PARTICIPANT FLOW:
Groups:
- TH-302 in Combination With Doxorubicin: 75 mg/m2 of Doxorubicin administered by bolus injection starting on Day 1 of a 21-day cycle.
  TH-302: TH-302 will be administered by IV infusion over 30-60 minutes on Days 1 and 8 of a 21-day cycle.
  Dose escalation dose levels:
  Dose level -1 (if needed): 180 mg/m2 Starting dose: 240 mg/m2
Period: Overall Study
Arm/Group | TH-302 in Combination With Doxorubicin
Started | 101
Completed All Treatment Cycles | 68
Completed | 68
Not Completed | 33

BASELINE CHARACTERISTICS:
Population: 107 enrolled, 101 dosed.
Arm/Group | TH-302 in Combination With Doxorubicin
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 77
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 86
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) Measured of TH-302 When Used in Combination With Doxorubicin and Prophylactic Growth Factor Support in Subjects With Advanced Soft Tissue Sarcoma
Time Frame: Two years
Measure: Number; unit: mg/m2
Arm/Group | TH-302 in Combination With Doxorubicin
Number analyzed (Participants) | 107
mg/m2 | 300

ADVERSE EVENTS:
Arm/Group | TH-302 in Combination With Doxorubicin
Serious Adverse Events (participants affected / at risk) | 64/101
Other Adverse Events (participants affected / at risk) | 101/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 in Combination With Doxorubicin (N=101)
Catheter site cellulitis (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1)
Infusion site infection (Infections and infestations) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1)
Neutropenic infection (Infections and infestations) | 2 (2)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Body temperature increased (Investigations) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 in Combination With Doxorubicin (N=101)
Urinary tract infection (Infections and infestations) | 16 (20)
Anaemia (Blood and lymphatic system disorders) | 72 (104)
Leukopenia (Blood and lymphatic system disorders) | 30 (85)
Neutropenia (Blood and lymphatic system disorders) | 31 (58)
Thrombocytopenia (Blood and lymphatic system disorders) | 53 (145)
Anorexia (Metabolism and nutrition disorders) | 40 (44)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11)
Dehydration (Metabolism and nutrition disorders) | 12 (13)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 28 (32)
Hypocalcaemia (Metabolism and nutrition disorders) | 12 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (28)
Hyponatraemia (Metabolism and nutrition disorders) | 13 (16)
Anxiety (Psychiatric disorders) | 11 (12)
Insomnia (Psychiatric disorders) | 12 (13)
Dizziness (Nervous system disorders) | 23 (25)
Dysgeusia (Nervous system disorders) | 17 (25)
Headache (Nervous system disorders) | 22 (30)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Abdominal pain (Gastrointestinal disorders) | 16 (16)
Constipation (Gastrointestinal disorders) | 46 (53)
Diarrhoea (Gastrointestinal disorders) | 37 (56)
Dyspepsia (Gastrointestinal disorders) | 13 (14)
Dysphagia (Gastrointestinal disorders) | 15 (16)
Haemorrhoids (Gastrointestinal disorders) | 17 (20)
Nausea (Gastrointestinal disorders) | 75 (110)
Stomatitis (Gastrointestinal disorders) | 49 (61)
Vomiting (Gastrointestinal disorders) | 36 (58)
Alopecia (Skin and subcutaneous tissue disorders) | 54 (55)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (32)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 (22)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 25 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (37)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (24)
Fatigue (General disorders) | 70 (83)
Oedema peripheral (General disorders) | 16 (22)
Pyrexia (General disorders) | 25 (33)
Blood alkaline phosphatase increased (Investigations) | 14 (14)
Weight decreased (Investigations) | 20 (20)
White blood cell count decreased (Investigations) | 13 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No